CLINICAL TRIAL: NCT00361452
Title: Acoustic Assessment of Nebulized Epinephrine Versus Albuterol for RSV Bronchiolitis- a Double Blind Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: epinephrine_albuterol_rsv.ctil
Record Dates: First submitted 2006-08-06; First posted 2006-08-08 (Estimated); Last update posted 2006-08-08 (Estimated); Status verified 2000-11

CONDITIONS: Rsv Bronchiolitis

INTERVENTIONS:
Drug: nebulized epinephrine and nebulized albuterol

SUMMARY:
Bronchiolitis is a common disease of infancy and a main reason for infants' hospital admissions in the first 2 years of life. The main cause of bronchiolitis is RSV (respiratory syncytial virus). Though, Treatment is mainly supportive, the treatment benefit of nebulized epinephrine or albuterol has been largely debated for the past years. Most of the clinical studies used clinical parameters to detect and compare the effectiveness of such medical interventions. In this study we will use non invasive computerized method of wheeze and crackles quantification to compare the effectiveness of nebulized epinephrine vs albuterol in RSV Bronchiolitis.

DETAILED DESCRIPTION:
Inpatient Infants younger than 2 years of age with first episode of RSV bronchiolitis will be randomly assigned to treatment with nebulized epinephrine (1 mg diluted with 3 ml of 0.9% saline) or nebulized albuterol (2.5 mg diluted with 3.5 ml of 0.9% saline). Both solutions will be provided in identical containers.

Clinical assessment and clinical score will be done before treatment, 10 and 30 minutes after treatment. The following parameters were recorded at each time point, wheezing, respiratory distress, O2 saturation, respiratory rate and heart rate. Computerized lung sounds as well, will be recorded before treatment, 10 and 30 minutes after treatment via 4 contact sensors attached to the chest.

ELIGIBILITY:
Inclusion Criteria:

* Under one year of age
* first episode of wheezing and dyspnea
* RSV antigen detected by ELISA
* parents signed informed consent.

Exclusion Criteria:

* infants with chronic lung disease
* cardiac disease
* other chronic conditions.

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30
Dates: Start 2000-12; Study Completion 2001-05

PRIMARY OUTCOMES:
respiratory clinical score
computerized quantification of wheezing and crackles

CONTACTS AND LOCATIONS:
Overall Officials: LEA BENTUR, MD, Principal Investigator — Rambam medical centre, pediatric pulmonary unit, HAIFA
Locations (1):
- Pediatric Ward, Rambam Medical Centre, Haifa, Israel

REFERENCES:
- [Derived] Beck R, Elias N, Shoval S, Tov N, Talmon G, Godfrey S, Bentur L. Computerized acoustic assessment of treatment efficacy of nebulized epinephrine and albuterol in RSV bronchiolitis. BMC Pediatr. 2007 Jun 2;7:22. doi: 10.1186/1471-2431-7-22. PMID 17543129